CLINICAL TRIAL: NCT05794581
Title: A Randomized, Double-Blind, Placebo and Comparator-Controlled Crossover Study to Assess the Effects of CT-868 Treatment on Glucose Homeostasis in Participants with Type 1 Diabetes
Brief Title: A Study to Assess the Effects of CT-868 Treatment on Glucose Homeostasis in Participants with Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Carmot Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-868-005
Record Dates: First submitted 2023-03-10; First posted 2023-04-03 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Obesity; Overweight
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Obesity; Overweight | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- CT-868 (Experimental): SC injection of CT-868 Intervention
  Interventions: Drug: CT-868
- Placebo (Placebo Comparator): SC injection of placebo matching CT-868 dose
  Interventions: Drug: Placebo
- Victoza (Active Comparator): SC injection of active comparator
  Interventions: Drug: Victoza

INTERVENTIONS:
Drug: CT-868 — CT-868
  Arms: CT-868
Drug: Placebo — Placebo as SC Injection
  Arms: Placebo
Drug: Victoza — Victoza as active comparator as SC Injection
  Other Names: Liraglutide
  Arms: Victoza

SUMMARY:
This study will be conducted primarily to evaluate the effects of CT-868 on glucose homeostasis in participants with Type 1 Diabetes Mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Female or male adults with Type 1 diabetes
* Ages 18-65 years
* Type 1 DM for at least 3 years
* Using an insulin pump or multiple daily injections (MDI) for at least 3 months
* BMI 25.0 - 35.0

Exclusion Criteria:

* Significant medical history
* Uncontrolled diabetes
* History of surgical treatment for weight loss
* History of malignancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2024-03-06 (Actual); Study Completion 2024-04-06 (Actual)

PRIMARY OUTCOMES:
To assess area under the curve (AUC) in glucose metabolism during MMTT | Baseline up to 4 days

SECONDARY OUTCOMES:
To assess changes in continuous glucose monitoring (CGM) measures | Baseline up to 4 days
Area under the acetaminophen concentration-time (AUC) | 0 - 300 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Carmot Clinical Research Unit 101, Chula Vista, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Carmot Therapeutics, Inc. — https://carmot-therapeutics.us/